CLINICAL TRIAL: NCT04693429
Title: Phase I Clinical Study for the Evaluation of Safety and Tolerability of PRO-172 Ophthalmic Solution, Manufactured by Laboratorios Sophia, S.A. de C.V., When Applied on the Ocular Surface of Healthy Volunteers
Brief Title: Clinical Study for the Evaluation of Safety and Tolerability of PRO-172 Ophthalmic Solution+
Acronym: PRO-172
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SOPH172-0919/I
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Safety; Tolerability; Ocular Surface; Ocular Comfort
MeSH Terms: interventions — bepotastine besilate

STUDY DESIGN:
Intervention Model Description: Controlled, single center, non comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRO-172 (Experimental): PRO-172 Ophthalmic Solution QID (four times per day). Single arm.
  Interventions: Drug: Bepotastine Besilate

INTERVENTIONS:
Drug: Bepotastine Besilate — Bepotastine Besilate 1.5% QID (quater in die) for 7 days
  Other Names: PRO-172

SUMMARY:
Clinical phase I, controlled, non comparative, open, single center study evaluating the safety and tolerability of ophthalmic solution PRO-172 when applied on the ocular surface of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy volunteers
* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Being between 18 and 45 years old.
* Women in child-bearing age must assure the continuation (start ≥ 30 days prior to informed consent signing) of a hormonal contraceptive method of intrauterine device (IUD) during the study.
* Having a best corrected visual acuity equal or better than 20/30 in both eyes.
* Showing normal vital signs.
* Having an intraocular pressure between 10 and 21 mmHg.

Exclusion Criteria:

* Using any kind of ophthalmic topical product.
* Using drugs or herbal products, through any administration route.
* For women: pregnancy, breastfeeding or planning to become pregnant during the time of the study.
* Having participated in clinical trials 90 days prior to inclusion in this study.
* Having participated previously in this study.
* Using contact lenses and not being able to suspend such use during the period of the study.
* Being unable to follow the lifestyle modification considerations required for the study.
* Having started the use of hormonal contraceptives of IUD within 30 days previous of inclusion in this study.
* Suffering any chronic degenerative diseases.
* Suffering active inflammatory of infectious disease when entering this study.
* Suffering unresolved lesions or traumas when entering this study.
* Having a previous history of any kind of ocular surgery.
* Having a previous history of any surgical procedure, non ophthalmological, within the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Clínica de Bioequivalencia, S. de R.L. de C.V., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRO-172
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Units Other Than Participants: Eyes
Arm/Group | PRO-172
Number analyzed (Participants) | 22
Number analyzed (Eyes) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.50 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 22
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmhg] | 13.75 (2.19)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Related Unexpected Adverse Events (AE)
Description: Presence/absence of related non expected adverse events
Time Frame: Day 10
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify adherence to stipulated procedures in the protocol.
Measure: Number; unit: Number of unexpected related AE
Arm/Group | PRO-172
Number analyzed (Participants) | 22
Number of unexpected related AE | 12

2. Primary Outcome: Ocular Comfort Index
Description: Ocular Comfort Index (OCI) Questionnaire for evaluation of dry eye symptoms in a scale from 0 to 100. Greater scores mean a worse outcome.
Time Frame: Day 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO-172
Number analyzed (Participants) | 22
score on a scale | 17.70 (11.76)

3. Secondary Outcome: Changes in Best Corrected Visual Acuity (BCVA)
Description: Visual acuity (VA) is a test of visual function. It will be evaluated with the Snellen chart. The Snellen chart is the standard tool used to evaluate visual acuity. It was located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20/20.This score can be expressed in fraction (i.e. 20/20) decimal (i.e. 1.0), or LogMAR (i.e. 0) formats. In this study, VA is expressed in decimal format. In decimal format, a lower number is a worse outcome.
Time Frame: Baseline vs Day 8
Measure: Mean (Standard Deviation); unit: decimal score (Snellen Chart)
Arm/Group | PRO-172
Number analyzed (Participants) | 22
decimal score (Snellen Chart) | 0.921 (0.125)

4. Secondary Outcome: Conjunctival and Corneal Staining With Lissamine Green
Description: Conjunctival and corneal staining with lissamine green. The evaluation will take place after applying the lissamine green stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V).
Time Frame: Day 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | PRO-172
Number analyzed (Participants) | 22
percentage of participants
  Oxford scale: Absent (0) | 60.5
  Oxford scale: Minimal (I) | 39.5

5. Secondary Outcome: Conjunctival and Corneal Staining With Fluorescein
Description: Conjunctival and corneal staining with fluorescein. The evaluation will take place after applying the fluorescein tain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V).
Time Frame: Day 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | PRO-172
Number analyzed (Participants) | 22
percentage of participants
  Oxford scale: Absent (0) | 81.6
  Oxford scale: Minimal (I) | 13.2
  Oxford scale: Mild (II) | 5.3

6. Secondary Outcome: Conjunctival Hyperemia
Description: Rate of conjunctival hyperemia will be evaluated through the Efron scale which includes 5 grades: Normal (0), Very Mild (I), Mild (II), Moderate (3), and Severe (4).
Time Frame: Day 8
Population: as for baseline characteristics
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | PRO-172
Number analyzed (Participants) | 22
Number analyzed (Eyes) | 44
percentage of eyes
  the Efron scale: Normal (0) | 60.5
  the Efron scale: Very Mild (I) | 39.5

7. Secondary Outcome: Chemosis Incidence
Description: Chemosis incidence will be evaluated at the end of the treatment at the final visit
Time Frame: Day 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-172
Number analyzed (Participants) | 22
Participants | 0

ADVERSE EVENTS:
Time Frame: From day 1 (basal visit) to the safety call on day 10 (± 1 days)
Description: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Arm/Group | PRO-172
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 17/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO-172 (N=22)
Irritation in the area of instillation (Eye disorders) | 7
Burning sensation (Eye disorders) | 11
Ocular discharge (Eye disorders) | 1
dysgeusia (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 1
pharyngitis (Gastrointestinal disorders) | 1
photophobia (Eye disorders) | 1
sore throat (Gastrointestinal disorders) | 1
heartburn (Gastrointestinal disorders) | 2
feeling of sticky eye (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04693429/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04693429/SAP_001.pdf